CLINICAL TRIAL: NCT01888770
Title: The Effect of Prematurity and Hypertensive Disorders of Pregnancy on Offspring Cardiovascular Health
Acronym: EPOCH
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Oxford (Other)
Collaborators: British Heart Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: EPOCH
Record Dates: First submitted 2013-06-13; First posted 2013-06-28 (Estimated); Last update posted 2016-05-25 (Estimated); Status verified 2016-05

CONDITIONS: Preeclampsia; Preterm Birth
MeSH Terms: conditions — Pre-Eclampsia; Premature Birth

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, serum, plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- Normotensive Term: Infants born at term (>37 weeks) to Normotensive pregnancies
- Term Preeclampsia: Infants born at term (>37 weeks gestation) and exposed to a preeclamptic pregnancy
- Preterm Normotensive: Infants born to Normotensive pregnancies at <37 weeks gestation
- Preterm Hypertensive: Infants born to hypertensive pregnancies at <37 weeks completed gestation
- Term Pregnancy-induced Hypertension: Infants born at term (>37 weeks gestation) and exposed to pregnancy-induced hypertension

SUMMARY:
The purpose of this study is to investigate whether exposure to hypertensive disorders of pregnancy and/or a preterm birth results in alterations in the cardiovascular system during infancy.

DETAILED DESCRIPTION:
While the incidence of cardiovascular disease has reduced dramatically, coinciding with favourable changes in risk factors, cardiovascular disease remains the single largest cause of mortality and premature mortality in the United Kingdom. Identification of novel biological pathways that underlie disease susceptibility raises the potential for new early primary prevention strategies to complement classical management. There is particular interest in the role of early environment in 'programming' risk of cardiovascular disease in later life and growing evidence that various early life exposures impact cardiovascular health in the longer term.

The investigators have therefore designed the EPOCH study to investigate whether those individuals born to hypertensive pregnancies and/or to a preterm birth demonstrate differences in the cardiovascular phenotype at birth, or whether they develop any differences over the first three months of life and whether this varies with other perinatal factors. This study also allows investigation of the short term impact of perinatal interventions used in this cohort. Comprehensive multi-modality non-invasive imaging measures of cardiovascular structure and function allow precise quantification of cardiovascular phenotype in this population.

ELIGIBILITY:
Inclusion Criteria:

* Available for assessment within the neonatal period,
* Parent is willing and able to give informed consent for participation in the study,
* Physical condition is suitable to allow non-invasive vascular testing,
* Mother meets criteria for inclusion in the study and is willing to participate in the study. (Aged >/= 16 years and Is able and willing to give informed consent for participation in the study, and is able and willing to give informed consent for her infants participation in the study. )
* Cases: Diagnosed during pregnancy with preeclampsia or gestational hypertension and/or delivered preterm (<37 weeks gestation)
* Controls: No history of gestational hypertension or preeclampsia during this pregnancy and delivered at term (>37 weeks gestation)

Exclusion Criteria:

* Parent is unwilling to give consent,
* Unavailable for assessment of cardiovascular system,
* Physical condition unsuitable to allow for non-invasive testing of cardiovascular system,
* Evidence of congenital cardiovascular disease (with the exception of Persistent Patent Ductus Arterious (PDA) and Atrial Septal Defect (ASD)),
* Cardiorespiratory instability at time of proposed measures,
* Active infection at time of proposed study measures,
* Mother of infant is excluded from the study. (Aged <16 years, unable or unwilling to consent to study or Physical condition post delivery such that it would preclude participation in the study)

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Study population is drawn from infants admitted to or delivered in the OUH NHS Foundation trust to normotensive or hypertensive pregnancies across a range of gestations. The mothers of these infants form a secondary study cohort.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2011-08; Primary Completion 2017-09 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Systolic Cardiac Function | Birth and 3 months
  Cardiac Function will be assessed by ECHO at birth and 3 months

SECONDARY OUTCOMES:
Micro-vascular Structure | Birth and 3 months
  Micro-vascular Structure will be assessed using Side Stream Dark Field (SDF) imaging device at birth and 3 months (as capillary density at baseline)
Pulse wave velocity and pulse-wave analysis | Birth and 3 months
Cardiac Structure | Birth and 3 months
  Cardiac structure will be assessed by echocardiography at in utero, at birth and 3 months (as left and right ventricular mass)
Cardiac diastolic function | Birth and 3 months
  Cardiac Function will be assessed by ECHO at birth and 3 months
Blood pressure | Birth and 3 months
Heart rate variability | Birth and 3 months
  Heart rate variability will be assessed by a 5 minute electrocardiogram

CONTACTS AND LOCATIONS:
Overall Officials: Paul Leeson, PhD, FRCP, Principal Investigator — University of Oxford Department of Cardiovascular Medicine
Locations (1):
- Cardiovascular Clinical Research Facility, Dept of Cardiovascular Medicine, University of Oxford, Oxford, Oxfordshire, United Kingdom